CLINICAL TRIAL: NCT06242002
Title: Early Post-operative Monitoring by Sensor of Patients Undergoing Forefoot Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique de lEurope a Amiens (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02074-41
Record Dates: First submitted 2024-01-25; First posted 2024-02-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Foot Injury
Keywords: foot; surgery; sensor; post-surgical follow-up
MeSH Terms: conditions — Foot Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): For patients participating to the clinical trial, the sensor will be positioned at the end of the procedure, under the surgical dressing, at ankle level.
  This dressing is a definitive dressing which is only removed during the post-operative consultation on day 8, during which the sensor will be removed.
  During this 7 days, data from the sensor will be collected every 4 hours.
  Interventions: Procedure: Set up of sensor

INTERVENTIONS:
Procedure: Set up of sensor — Surgery is performed as usual for patients needing this medical procedure. At the end, the sensor is set up under the surgical dressing.

SUMMARY:
The goal of this clinical trial is to evaluate the monitoring using a sensor in patients who have undergone forefoot surgery, during the first 7 post-operative days.

The monitoring tool has a Global Positioning System (GPS) beacon, a 3-axis accelerometer and a temperature sensor, as well as an "emergency call" button.

The main objective it aims to answer are:

* to evaluate the feasibility of post-operative monitoring using this tool
* to evaluate the reliability of the tool

The investigators hope to determine if using this tool can be able to provide patients a "connected" personalized real-time monitoring for follow-up.

DETAILED DESCRIPTION:
Currently, patients undergoing forefoot surgery often do so in an outpatient setting and thus spend less and less time in the healthcare establishment in contact with the nursing staff, being increasingly left to themselves at home. The development of telemedicine with real-time information transfer can enable the monitoring of acute or chronic pathologies, thus allowing a link between the patient and the healthcare network, for more personalized monitoring.

Post-operative pain following forefoot surgery is now well controlled, allowing greater patient autonomy despite post-operative footwear. However, the patient's autonomy, locomotor and mobilization capacity are not known.

The investigators therefore propose monitoring the first 7 post-operative days using a sensor in patients who have undergone forefoot surgery. This 7-day period corresponds to the critical period of foot surgery with resumption of post-operative support, lifting of loco-regional anesthesia and return home. This monitoring will be done from discharge from the service until the first post-operative visit. The monitoring will be prospective with non-invasive measurements via an electronic sensor (already used for sporting activities, notably long-distance running). This will be a clinical practice study, with no modification to monitoring or current practices. The monitoring tool has a Global Positioning System (GPS) beacon, a 3-axis accelerometer and a temperature sensor, as well as an "emergency call" button. The recorded parameters will be the number of steps, local temperature and GPS position of the patient. The data will be transmitted via an independent cellular network and to a secure space (username and password) accessible online.

The main objective will be to evaluate the feasibility of post-operative monitoring using this tool. The secondary objectives will be to evaluate the reliability of the tool, to evaluate the transmission of the GPS signal, and to collect the data.

Following this study, the investigators hope to be able to provide patients with real-time monitoring, via alerts received on the smartphone (e.g. icing instructions via the temperature sensor, instructions to reduce locomotor activity, etc.) .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing forefoot surgery
* Patient having given informed consent

Exclusion Criteria:

* Patient deprived of his liberty or under guardianship
* Patient undergoing surgery other than the forefoot (hallux and lateral toes)
* Patient unable to undergo protocol monitoring for psychological, social, family, geographic or linguistic reasons
* Patient with an underlying or concomitant pathology incompatible with inclusion in the trial, whether psychiatric or somatic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Step count | Every 4 hours during 7 days
  Collecting step count data on the server
local temperature | Every 4 hours during 7 days
  Collecting local temperature data on the server
distance traveled (kilometers) | Every 4 hours during 7 days
  Collecting data on the distance traveled by the patient on the server, (in kilometers). Distance is measured by the global positioning system beacon of the sensor.

SECONDARY OUTCOMES:
Patient's satisfaction : questionnaire | day 8
  Patients satisfaction will be evaluated by a questionnaire with 5 items. 4 items are "yes-no" questions, and the last one is a Likert scale of 5 levels (from "not at all satisfied" to "very satisfied").

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de l'Europe à Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No